CLINICAL TRIAL: NCT00476580
Title: Health Habits and Cancer Risk Among a US Migrant Sri Lankan Population and a Comparison With Siblings Living in Sri Lanka
Brief Title: Health Habits and Cancer Risk Comparison Among Migrant Sri Lankans and Sri Lankans
Status: Withdrawn | Type: Observational
Why Stopped: Study terminated.
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 2006-1047
Record Dates: First submitted 2007-05-21; First posted 2007-05-22 (Estimated); Last update posted 2015-08-28 (Estimated); Status verified 2015-08

CONDITIONS: Acculturation
Keywords: Sri Lankan Sinhalese; Epidemiology; Cancer Risk; US Migrant; Questionnaire; Survey; Acculturation; Health and Cancer Risks; Health Habits
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Sri Lankan Sinhalese: Sri Lankan Sinhalese adults (18 years of age or older) living in the greater Houston area, but born in Sri Lanka.
  Interventions: Behavioral: Questionnaire
- Siblings or Cousins in Sri Lanka: Siblings or the first cousins of the study participants living in Sri Lanka of same sex and of an age plus or minus 10 years.
  Interventions: Behavioral: Questionnaire

INTERVENTIONS:
Behavioral: Questionnaire — Questions to collect health information specific to Sri Lankans.
  Other Names: Survey

SUMMARY:
Objectives:

General objective:

To determine how acculturation to United States has influenced the health and cancer risk among a US migrant Sri Lankan population.

Specific objectives:

1. To determine the prevalence of cancer and cancer related non-communicable diseases among Sri Lankan Sinhalese living in the greater Houston area.
2. To study the distribution of risk factors for cancer in this population.
3. To study the pattern of utilization of methods available for early detection of cancer in this population.
4. To study and compare the findings of this survey with that of the siblings of this population living in Sri Lanka.

DETAILED DESCRIPTION:
A health survey among Sinhala adults living in Houston comparing the health and health habits between the Sri Lankans living in Houston and their close relatives living in Sri Lanka.

ELIGIBILITY:
Inclusion Criteria:

1. Sri Lankan Sinhalese adults (18 years of age or older) living in the greater Houston area but born in Sri Lanka
2. Siblings or the first cousins of the study participants living in Sri Lanka of same sex and of an age plus or minus 10 years

Exclusion Criteria:

1. Sri Lankan Sinhalese born in the US
2. Sri Lankan Sinhalese under 18 years of age
3. Participation in a M. D. Anderson sponsored focus group or survey regarding health within the past 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Sri Lankan Sinhalese adults (18 years of age or older) living in the greater Houston area, but born in Sri Lanka. Siblings or the first cousins of the study participants living in Sri Lanka of same sex and of an age plus or minus 10 years.
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2007-04; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Determine how acculturation to US has influenced health and cancer risk (prevalence of cancer related non-communicable diseases, distribution of risk factors, early cancer detection method utilization) among Sri Lankan Sinhalese in greater Houston area. | 3 Years

SECONDARY OUTCOMES:
To study and compare the findings of this survey with that of the siblings of this population living in Sri Lanka. | 1 Year

CONTACTS AND LOCATIONS:
Overall Officials: Richard A. Hajek, PHD, MS, BA, Principal Investigator — M.D. Anderson Cancer Center
Locations (3):
- United States (2):
  - University of Texas MD Anderson Cancer Center, Houston, Texas
  - City of Houston Department of Health and Human Services, Houston, Texas
- University of Peradeniya, Peradeniya, Sri Lanka

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org